CLINICAL TRIAL: NCT02080403
Title: Multi-Center Phase 3 Trial of Chlorhexidine Gluconate Chip for the Use in Subjects With Peri-Implantitis.
Brief Title: The Efficacy and Safety of Chlorhexidine Gluconate Chip (PerioChip®) in Therapy of Peri-implantitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexcel Pharma Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLI/016P
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis; Periodontal Diseases; Chlorhexidine gluconate; PerioChip; Anti-Infective Agents; Mouth Diseases; Antiseptics
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases; Mouth Diseases | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Treatment, 2.5 mg Chlorhexidine Gluconate chip (PerioChip®) inserted every two weeks starting at Baseline for the first 3 months, plus mechanical Subgingival Debridement at Baseline and 3 months.
  Interventions: Drug: 2.5 mg Chlorhexidine gluconate chip
- Control (No Intervention): Mechanical Subgingival Debridement at Baseline and 3 months.

INTERVENTIONS:
Drug: 2.5 mg Chlorhexidine gluconate chip — Subgingival debridement will be carried out for each one of the target implant. Upon completion of the debridement a PerioChip® will be inserted in each one of the target implant.
  Other Names: PerioChip®
  Arms: Treatment

SUMMARY:
The objective of the study is to assess the efficacy and safety of PerioChip® (Chlorhexidine gluconate chip) in the treatment of patients with Peri-implantitis.

The hypothesis of the study is that PerioChip® in adjunct to mechanical subgingival debridement is more effective in the treatment of peri-implantitis when compared to the common method of mechanical subgingival debridement alone. The primary efficacy measure will be the reduction in probing pocket depth at 6 months as measured at sites of qualifying target implant.

DETAILED DESCRIPTION:
This is a research study that uses the drug PerioChip® (active ingredient chlorhexidine gluconate) as an experimental treatment for "periimplantitis". This condition is defined an inflammation affecting the tissues (gums and bone) around an already stable implant, resulting in loss of supporting jaw bone. It is caused by many factors but current research links the condition with the presence of bacteria in the mouth which are responsible for periodontitis (gum disease). If left untreated, this can lead to decreased bone support, weakening of the implant and potential lost of the implant.

Nonsurgical treatment (deep cleaning with instruments to remove plaque) and rigorous diligent oral care at home are commonly used to treat both periimplantitis (gum disease around an implant) and periodontitis (gum disease around teeth).

The medication PerioChip® is a small dental chip (its size is smaller than a match head, and it is completely flat). The chip contains chlorhexidine gluconate, an antimicrobial agent which is not an antibiotic. The chip is inserted into the gum sulcus that is present around the tooth or implant and biodegrades naturally within 7 to 10 days while releasing the medication.

The purpose of this study is to determine the efficacy of PerioChip® in addition to a standard deep cleaning treatment regime, as compared to standard deep cleaning alone.in a large patient population, and to collect additional safety data about the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* At least one implant in the oral cavity with clinical and radiographical signs of peri-implantitis. Including bone loss in combination with bleeding and/or suppuration on probing and a peri-implant Probing Depth (PD) of 5-8 mm.
* The implants have been in function for more than 2 years.
* Fixed prosthetic restoration of the implant.

Exclusion Criteria:

* Pregnancy.
* Patient uses Chlorhexidine oral rinses/ mouthwashes on a regular basis.
* Allergic reaction to Chlorhexidine.
* Active Periodontitis which required definitive treatment.
* Presence of orthodontic appliances, or any removable appliances, that impinges on the tissues being assessed.
* Use of systemic antibiotic therapy and/or chronically use of non-steroidal anti-inflammatory drugs (NSAIDs).
* Uncontrolled diabetes, of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Machtei, Prof., Study Chair — Department of Periodontology, School of Graduate Dentistry, Rambam Health Care Center Haifa, Israel, 9602
Locations (10):
- United States (6):
  - University of Maryland, School of Dentistry, Department of Periodontics, Baltimore, Maryland
  - The Harvard School of Dental Medicine, Boston, Massachusetts
  - Tufts University, School of Dental Medicine, Department of Oral Medicine, Boston, Massachusetts
  - University of Michigan, School of Dentistry, Department of Periodontics and Oral Medicine, Ann Arbor, Michigan
  - Columbia University, College of Dental Medicine ,Division of Periodontics, New York, New York
  - Stony Brook University, School of Dental Medicine, Department of Periodontology, Stony Brook, New York
- Zentrum für Zahn,- Mund- und Kieferheilkunde Poliklinik für Parodontologie, Giessen, Germany
- Israel (2):
  - Department of Periodontology, School of Graduate Dentistry, Rambam Health Care Center, Haifa
  - The Faculty of Dental Medicine, Department of Periodontics, Hadassah Ein Karem, Jerusalem
- Institute of Dentistry, Barts & The London School of Medicine & Dentistry, Queen Mary University of London (QMUL), London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 146 | 144
Completed | 131 | 132
Not Completed | 15 | 12
Not completed — Adverse Event | 5 | 1
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 3 | 7
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 146 | 144 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.2) | 62.6 (11.6) | 62.6 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 81 | 172
  Male | 55 | 63 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 9 | 23
  Not Hispanic or Latino | 131 | 134 | 265
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 3 | 13
  White | 117 | 127 | 244
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 95 | 93 | 188
  United Kingdom | 10 | 11 | 21
  Israel | 30 | 28 | 58
  Germany | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Probing Pocket Depth for Selected Target Implants
Description: Pocket depth was measured as the distance from the coronal edge of the gingival margin to the base of the pocket. It was assessed at 4 sites per implant: mesiobuccal, midbuccal, distobuccal, and midlingual. Only one of the 4 sites, usually the deepest, was determine to be target implant.
Time Frame: Baseline to 6 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target implant
Arm/Group | Treatment | Control
Number analyzed (Participants) | 146 | 144
Number analyzed (Target implant) | 180 | 174
mm | -1.69 (1.18) | -1.51 (1.16)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.1159, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.40 to 0.04]

2. Secondary Outcome: Absolute Change in Mean Probing Pocket Depth of Selected Target Implants in Patients With Baseline Pocket Depth Measurement of 6-8 mm Inclusive
Description: as for outcome 1
Time Frame: Baseline to 6 months
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target implant
Arm/Group | Treatment | Control
Number analyzed (Participants) | 146 | 144
Number analyzed (Target implant) | 141 | 130
mm | -1.77 (1.25) | -1.65 (1.18)

3. Secondary Outcome: Percentage of Selected Target Implants Bleeding on Probing (BOP)
Description: The proportion of the change in bleeding status (bleeding to no bleeding) for the selected target implant
Time Frame: 6 months
Population: Intent to Treat
Measure: Count of Units; unit: Target implant
Units Other Than Participants: Target implant
Arm/Group | Treatment | Control
Number analyzed (Participants) | 146 | 144
Number analyzed (Target implant) | 180 | 173
Target implant | 90 | 77

4. Secondary Outcome: Precentage of Selected Target Implant BOP
Description: The proportion of change in bleeding status (bleeding to no bleeding) for selected target implant
Time Frame: Week 16
Measure: Count of Units; unit: Target implant
Units Other Than Participants: Target implant
Arm/Group | Treatment | Control
Number analyzed (Participants) | 146 | 144
Number analyzed (Target implant) | 179 | 165
Target implant | 76 | 73

ADVERSE EVENTS:
Time Frame: Screening through Week 24
Description: All randomized patients who were treated with at least 1 study treatment or who underwent subgingival debridement.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/146 | 2/144
Serious Adverse Events (participants affected / at risk) | 4/146 | 3/144
Other Adverse Events (participants affected / at risk) | 43/146 | 19/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=146) | Control (N=144)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Forearm fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=146) | Control (N=144)
Implant site pain (General disorders) | 12 | 0
Nasopharyngitis (Infections and infestations) | 5 | 7
Post procedural discomfort (Injury, poisoning and procedural complications) | 5 | 1
Tooth repair (Surgical and medical procedures) | 3 | 2
Aphthous ulcer (Gastrointestinal disorders) | 3 | 1
Gingivitis (Infections and infestations) | 1 | 3
Toothache (Gastrointestinal disorders) | 5 | 0
Artificial crown procedure (Surgical and medical procedures) | 3 | 0
Gingival pain (Gastrointestinal disorders) | 3 | 0
Headache (Nervous system disorders) | 0 | 4
Implant site swelling (General disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Version 7 (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT02080403/Prot_000.pdf
  • Study Protocol: Version 8 (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT02080403/Prot_001.pdf
  • Study Protocol: Summary of Protocol Changes (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT02080403/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT02080403/SAP_003.pdf